CLINICAL TRIAL: NCT02301442
Title: A Randomised Controlled Trial of an Exercise Plus Behaviour Change Intervention in People With MS: the "Step it Up" Study Protocol
Brief Title: Step it Up: An Exercise and Behaviour Change Programme for People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ULimerick
Record Dates: First submitted 2014-11-13; First posted 2014-11-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise + behaviour change intervention (Experimental): This arm of the trial includes assessments at weeks 0, 12, 24 and 36. A 10-week exercise + behaviour change intervention will be delivered by physiotherapists between weeks 1 and 11.
  Interventions: Behavioral: Exercise + behaviour change intervention
- Exercise + control education (Active Comparator): This arm of the trial includes assessments at weeks 0, 12, 24 and 36. A 10-week exercise + control education intervention will be delivered by physiotherapists between weeks 1 and 11.
  Interventions: Behavioral: Exercise + control education

INTERVENTIONS:
Behavioral: Exercise + behaviour change intervention — In addition to the same exercise intervention as the control group, this group will receive a behaviour change intervention. This will be delivered after each exercise session and will incorporate the elements: self-efficacy, outcome expectations, impediments and goal-setting. On the weeks when the participants do not attend group sessions, they will receive telephone calls from physiotherapists. This will consist of guided conversations that consider content delivered in previous sessions.
  Arms: Exercise + behaviour change intervention
Behavioral: Exercise + control education — The control group will receive exercise and education components. The exercise intervention includes aerobic & strengthening components and are in line with MS exercise guidelines (Latimer-Cheung et al 2013). The aerobic activity is walking, measured using pedometers & exercise logs. The strengthening programme consists of 10 exercises targeting major muscle groups for the upper and lower extremities using elastic resistance band. Over the 10-week programme participants will attend 6 group exercise class, supplemented with telephone calls in the weeks without classes. After each group exercise class this group will receive an education session about the following: diet, vitamin D, sleep, temperature and hydration, and immunisations and vaccinations.
  Arms: Exercise + control education

SUMMARY:
Exercise has consistently yielded short-term, positive effects on health outcomes in people with multiple sclerosis (MS). However, these effects have not been maintained in the long-term. Behaviour change interventions aim to promote long-term positive lifestyle change. This study, namely, "Step it Up" will compare the effectiveness of an exercise plus Social Cognitive Theory (SCT)-based behaviour change intervention with an exercise plus control education intervention on walking mobility among people with MS.

DETAILED DESCRIPTION:
1. Background and study aims Exercise has consistently yielded short-term, positive effects on health outcomes in people with multiple sclerosis (MS). However, these effects have not been maintained in the long-term. Behaviour change interventions aim to promote long-term positive lifestyle change. This study, namely, "Step it Up" will compare the effect of an exercise plus Social Cognitive Theory (SCT)-based behaviour change intervention with an exercise plus control education intervention on walking mobility among people with MS. Our hypothesis is that those in the exercise and SCT-based intervention will achieve significantly more improvement in walking mobility than the control group post-intervention (12 weeks) and that this improvement will be maintained at 24- and 36- week follow up.
2. What does the study involve? Exercise plus contact control education intervention The control group will receive an exercise and a didactic control education component. The exercise intervention will include aerobic and strengthening components and will be delivered by physiotherapists. The aim of the exercise component is to progressively increase the intensity of both aerobic and strengthening activities to enable the participants to reach the recently published MS exercise guidelines (Latimer- Cheung et al 2013). The aerobic activity will be walking, the intensity of which will be monitored using step rate measured using the Yamax digiwalker pedometer* (which will be provided to all participants) and an exercise log to document duration of walking exercise and number of steps taken. It is widely accepted that 100 steps per minute equates to three MET or moderate intensity physically active (PA) among people with MS (Agiovlasitis and Motl 2014). Participants will begin with 10 minutes of walking twice weekly at a rate of 100 steps/minute and increase incrementally in 5 minute intervals over 5 weeks until they reach the guideline of 30 minutes twice weekly (Latimer-Cheung et al 2013).

The strengthening programme is based on a community-based exercise programme that has been evaluated previously (Garrett et al 2013) and will consist of 10 exercises targeting major muscle groups for the upper and lower extremities using elastic resistance band. Participants will begin with one set of 10-15 repetitions and gradually increase the number of sets, repetitions and level of resistance until they meet the target of two sets of each exercise twice weekly with sufficient resistance that they are failing on the 12th repetition. Over the 10-week programme participants will attend the group exercise class on six occasions, supplemented with a telephone coaching call in the weeks without classes (intervention weeks 4, 6, 7 and 9). These telephone calls will consist of direct questions about the frequency, intensity, type and duration of exercise they have completed and whether they have experienced any adverse events or relapses. After each of the group exercise classes the control group will receive an education session about topics unrelated to physical activity behaviour, e.g. diet, vitamin D, sleep, temperature and hydration, and immunisations and vaccinations.

Exercise plus SCT-based intervention The exercise plus SCT-based intervention group will receive the same exercise intervention as the control group (as described in the previous section).This group will also receive a behaviour change intervention based on the principles of SCT. The SCT-based education sessions will be delivered after each exercise session by physiotherapists and will incorporate the principle elements of SCT including self-efficacy, outcome expectations, impediments and goal-setting. Beyond providing presentation notes, individual reflection and written exercises, group discussion on each of the principles of SCT, and providing on-going feedback on all aspects of PA behaviour, the program will include video files of people with MS discussing PA behaviour and their experiences of initiating and maintaining a physically-active lifestyle. On the weeks when the participants do not attend group sessions, they will receive a telephone coaching call from the physiotherapist. These coaching calls will consist of guided conversations that consider the components of SCT delivered in the previous session and a revision of other components.

4. What are the possible benefits and risks of participating? Benefits to the participants include access to a free physiotherapy-led exercise programme, of which benefits such as improved aerobic capacity, mobility, fatigue, mood, muscle strength are anticipated. The education session may also help participants to keep those benefits for longer. The investigators do not envisage any adverse effects of these interventions.

5. Where is the study run from? This study has been organised by Clinical Therapies, University of Limerick.

6. When is study starting and how long is it expected to run for? This study started in September 2014 and it is anticipated that data collection will end in March 2016. Participants will be recruited until June 2015.

7. Who is funding the study? The Irish Health Research Board, Health Research Award Grant is funding the study.

8. Who is the main contact? Dr. Susan Coote (susan.coote@ul.ie)

ELIGIBILITY:
Inclusion Criteria:

* Physician-confirmed formal diagnosis of MS
* Patient Determined Disease Steps score of 0-3
* A sedentary lifestyle (< 30 minutes of moderate to strenuous exercise one day or more per week over the last six months)
* Willing to give written informed consent.

Exclusion Criteria:

* Pregnancy
* MS relapse in the last 12 weeks
* Changes to MS medication or steroid treatment in the last 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in walking mobility from weeks 1 to 36 | Weeks 1 to 36
  Change in walking mobility will be measured using the Timed up and Go test, the Six Minute Walk Test and the Multiple Sclerosis Walking Scale-12. These measures will be completed at weeks 1, 12, 24 and 36. The primary outcome will be the change over time from week 1 to week 36.

SECONDARY OUTCOMES:
Change in lower limb functional muscle strength from weeks 1 to 36 | Weeks 1 to 36
  Change in lower limb muscle strength will be measured using the 5 times sit to stand test. This measure will be completed at weeks 1, 12, 24 and 36.
Change in aerobic fitness from weeks 1 to 36 | Weeks 1 to 36
  Change in aerobic fitness will be measured using the Modified Canadian Aerobic Fitness Test. This measure will be completed at weeks 1, 12, 24 and 36.
Change in anxiety and depression from weeks 1 to 36 | Weeks 1 to 36
  Change in anxiety and depression will be measured using the Hospital Anxiety and Depression Scale. This measure will be completed at weeks 1, 12, 24 and 36.
Change in cognitive processing from weeks 1 to 36 | Weeks 1 to 36
  Change in cognitive processing will be measured using the Symbol Digit Modalities Test. This measure will be completed at weeks 1, 12, 24 and 36.
Change in physical activity levels from weeks 1 to 36 | Weeks 1 to 36
  Change in phyiscal activity levels will be measured using the Godin Leisure-Time Exercise Questionnaire, the International Physical Activity Questionnaire and an objective measure of physical activity- the SenseWear Arm band accelerometer. These measures will be completed at weeks 1, 12, 24 and 36.
Change in self-reported fatigue from weeks 1 to 36 | Weeks 1 to 36
  Change in self-reported fatigue will be measured using the Modified Fatigue Impact Scale. This measure will be completed at weeks 1, 12, 24 and 36.
Change in self-reported impact of MS from weeks 1 to 36 | Weeks 1 to 36
  Change in self-reported impact of MS will be measured using the Multiple Sclerosis Impact Scale-29. This measure will be completed at weeks 1, 12, 24 and 36.

OTHER OUTCOMES:
Adherence to the intervention | Week 12
  Participants adherence to the intervention will be measured at week 12 (post-intervention) using self-report (participant-reported) exercise logs and adherence logs recorded by the trial interventionalists.
Change in Social Cognitive Theory domains from weeks 1 to 36 | Weeks 1 to 36
  Change in Social Cognitive Theory domains will be measured using the Exercise Self-Efficacy Scale, the Exercise Goal Setting scale, the Multidimensional Outcomes Expectations for Exercise Scale and the Social Provisions Scale. These measures will be completed at weeks 1, 12, 24 and 36.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Coote, PhD, Principal Investigator — University of Limerick
Locations (1):
- Department of Clinical Therapies, University of Limerick, Limerick, Munster, Ireland

REFERENCES:
- [Derived] Hayes S, Uszynski MK, Motl RW, Gallagher S, Larkin A, Newell J, Scarrott C, Coote S. Randomised controlled pilot trial of an exercise plus behaviour change intervention in people with multiple sclerosis: the Step it Up study. BMJ Open. 2017 Oct 12;7(10):e016336. doi: 10.1136/bmjopen-2017-016336. PMID 29025830
- [Derived] Coote S, Uszynski M, Herring MP, Hayes S, Scarrott C, Newell J, Gallagher S, Larkin A, Motl RW. Effect of exercising at minimum recommendations of the multiple sclerosis exercise guideline combined with structured education or attention control education - secondary results of the step it up randomised controlled trial. BMC Neurol. 2017 Jun 24;17(1):119. doi: 10.1186/s12883-017-0898-y. PMID 28646860
- [Derived] Coote S, Gallagher S, Msetfi R, Larkin A, Newell J, Motl RW, Hayes S. A randomised controlled trial of an exercise plus behaviour change intervention in people with multiple sclerosis: the step it up study protocol. BMC Neurol. 2014 Dec 21;14:241. doi: 10.1186/s12883-014-0241-9. PMID 25528262